CLINICAL TRIAL: NCT02921126
Title: Real-World Evidence of Anticoagulation Treatment In Non-Valvular Atrial Fibrillation In Italy
Acronym: RE-FIT
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-494
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Anticoagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- High Dose Group: Apixaban - 10 mg/day Rivaroxaban - 20 mg/day Dabigatran - 300 mg/day
- Low Dose Group: Apixaban - 5 mg/day Rivaroxaban - 15 mg/day Dabigatran - 220 mg/day
- Other Dose Group: Invalid Doses / Off-Label

SUMMARY:
To quantify rates of bleeding events and investigate the characteristics of prescribed patients, rates of bleeding events, persistence and healthcare resource utilization of Oral Anticoagulants (OACs) prescribed in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* are at least 18 years of age at index date
* Initiated new OAC therapy ( no previous prescriptions of the same index OAC in the last 12 months prior to the index date ) during the study period
* Had at least 1 claim with diagnosis of AF anytime in their records

Exclusion Criteria:

* Have a record that is indicative of Valvular Atrial Fibrillation during this period
* Have a history of the OACs prescribed during the study period as assessed during the period of data availability(i.e. history of index OAC, as patients need to be newly prescribed either apixaban, rivaroxaban, dabigatran or VKA)
* Have more than one OAC exposure which starts on the same date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adults with NVAF who are newly prescribed apixaban, rivaroxaban, dabigatran, and VKA in 10 Italian Local Health Units (LHUs), during the study period, and meet the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 9914 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically relevant bleeding events among Non-valvular atrial fibrillation (NVAF) patients following treatment initiation on an oral OAC in Italy | Approximately 30 months

SECONDARY OUTCOMES:
Distribution of patient demographics at the time of OAC initiation | at baseline
Distribution of clinical characteristics at the time of OAC initiation | at baseline
Composite of number and percentage of patients who are persistent with their newly prescribed OAC | Approximately 30 months
Incidence of major bleeding events following treatment initiation among NVAF patients following treatment initiation on an oral OAC in Italy | Approximately 30 months
Composite of number and percentage of patients with major bleeding events, thromboembolic events, or death while exposed to the newly prescribed OAC | Approximately 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Ravenna, Italy

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx